CLINICAL TRIAL: NCT00192387
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial to Investigate Viral Shedding in Healthy Children (6 Mos and Less Than or Equal to 18 Months of Age) Vaccinated With Two Doses of Liquid Formulation of Influenza Virus Vaccine, Live Cold Adapted (CAIV-T)
Brief Title: Trial to Investigate Viral Shedding in Healthy Children Vaccinated With Vaccine Virus Liquid (CAIV-T)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: D153-P005
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2006-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Fluid Therapy

INTERVENTIONS:
Biological: CAIV-T, Liquid

SUMMARY:
The primary objective of this study was to determine the proportion of subjects, seronegative to all three strains of influenza, as defined by a serum hemagglutination inhibition antibodies (HAI) antibody titer of <1:10, who shed each vaccine virus strain following a single dose of CAIV-T.

ELIGIBILITY:
Inclusion Criteria:

* children at least 6 months of age and less than or equal to 18 months of age at the time of enrollment, and in good health as determined by medical history, physical examination, and clinical judgment;
* whose parent/legal guardian has provided written informed consent after the nature of the study has been explained;
* who, along with their parent or legal guardian, will be available for the two month duration of the trial (from enrollment to study completion).

Exclusion Criteria:

* whose parents or legal guardians are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids; intranasal steroids or cytotoxic agents;
* have an immunosuppressed or an immunocompromised individual living in the same household;
* with a documented history of hypersensitivity to egg or egg protein or any other component of the study vaccine or placebo;
* who, at anytime prior to study enrollment, receives any influenza vaccine (commercial or investigational);
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results.

Note: A pregnant household member is not considered a contraindication to enrollment.

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2001-09; Study Completion 2001-12

PRIMARY OUTCOMES:
Measurement of influenza-specific immune response following receipt of CAIV-T.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (1):
- Monroe Clinic, Monroe, Wisconsin, United States